CLINICAL TRIAL: NCT05184478
Title: A Pilot Randomized Placebo-controlled Crossover Trial of Medicinal Cannabis (MC) in Adolescents with Tourette Syndrome (TS)
Brief Title: Is Medicinal Cannabis an Effective Treatment for Tourette Syndrome in Adolescents? a Pilot Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RCH HREC 69238
Record Dates: First submitted 2021-12-02; First posted 2022-01-11 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-04

CONDITIONS: Tourette Syndrome in Adolescence
MeSH Terms: interventions — Medical Marijuana

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized 1:1 to initially receive either THC:CBD 10:15 oil or placebo in Treatment Period 1, before crossing over and receiving the other study drug (THC:CBD 10:15 oil or placebo) in Treatment Period 2.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (MC then placebo) (Experimental): Group A will receive medicinal cannabis during Treatment Period 1 (70 days), followed by a 7 day dose reduction and 21 day wash-out period, then will receive placebo during Treatment Period 2 (70 days).
  Interventions: Drug: Medicinal cannabis (MC): THC 10mg/mL : CBD 15mg/mL, manufactured by Cann Group Ltd.; Drug: Placebo
- Group B (placebo then MC) (Experimental): Group B will receive placebo during Treatment Period 1 (70 days), followed by a 7 day dose reduction and 21 day wash-out period, then will receive medicinal cannabis during Treatment Period 2 (70 days).
  Interventions: Drug: Medicinal cannabis (MC): THC 10mg/mL : CBD 15mg/mL, manufactured by Cann Group Ltd.; Drug: Placebo

INTERVENTIONS:
Drug: Medicinal cannabis (MC): THC 10mg/mL : CBD 15mg/mL, manufactured by Cann Group Ltd. — Each 1mL contains 10mg tetrahydrocannabinol (THC),15 mg cannabidiol (CBD), and 0.004mL peppermint oil in medium chain triglyceride (MCT) oil.
  All participants will start at 0.1 mL per day, and will gradually increase in 0.1mL increments until day 21 when a dose of 0.5mL (participants weighing <50kg) or 1mL (participants weighing ≥50kg) is reached. At day 29, an assessment of treatment response will be conducted. Participants who meet criteria for a treatment response will remain on the same dose for the remainder of the treatment period. Participants who do not meet criteria for a treatment response will gradually increase the dose in 0.1mL increments until day 49 when a daily dose of 1mL (participants weighing <50kg) or 2mL (participants ≥50kg) is reached.
Drug: Placebo — The placebo contains MCT oil and peppermint flavoring solution, which is indistinguishable from the active medication in appearance, smell and taste.
  The dose will be matched for volume to the medicinal cannabis, and will follow the same dosing schedule as the medicinal cannabis treatment phase.

SUMMARY:
This is a single site, pilot double-blind, randomized, placebo-controlled, cross-over study of 10 participants comparing medicinal cannabis (THC:CBD 10:15 oil) with placebo in reducing tics in adolescents aged 12 - 18 years with severe Tourette Syndrome (TS).

The primary objective of this pilot study is to evaluate all elements of the study design (recruitment strategy, study duration, study procedures, study medication tolerance and outcome measures) to assess if they are acceptable and feasible for the conduct of a full-scale randomized controlled trial of THC:CBD 10:15 oil to reduce tic severity in adolescents with TS.

The secondary objective of this study is to collect preliminary data on the safety of oral THC:CBD 10:15 oil in adolescents aged 12 to 18 years with TS.

As an exploratory aim data from clinician- and parent-rated measures will be compared across the phases to explore for a signal of efficacy on primary (tic reduction) and secondary (premonitory urges, obsessive compulsive behaviors, Attention Deficit Hyperactivity Disorder [ADHD] symptoms) outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 12 - 18 years of age;
* DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition) diagnosis of TS as assessed by the study clinician;
* TS severity defined as a score of 20 or higher on the Total Tic Severity section of the Yale Global Tic Severity Scale;
* No changes in either medication or other interventions in the 4 weeks prior to randomization, and intention to remain on same dose for the duration of the study;
* Participant and family have the ability to comply with the protocol requirements, in the opinion of the investigator;
* Agrees not to drive for the duration of the study.

Exclusion Criteria:

* Non-English speaking parents;
* Participant history of psychosis, schizophrenia, bipolar disorder, or major depressive disorder, or a family history of psychosis;
* Taking anti-epileptic medications which interact with medicinal cannabis: clobazam, mTOR (mammalian target of rapamycin) inhibitors (e.g sirolimus, tacrolimus), anti-cancer agents, citalopram >20mg/day, escitalopram >10mg/day;
* Abnormal liver function tests defined as ALT (alanine transaminase) > twice ULN (upper limit of normal);
* Current use of illicit drugs or medicinal cannabis, or use in the 4 weeks prior to screening;
* Pregnant or intending to become pregnant during the study, or breastfeeding;
* History of clinically significant suicidal thoughts in the prior 12 months.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Rate of study participant recruitment, calculated as the time required to reach a sample size of 10. | From the date of pre-screening the first participant until the tenth participant is randomized, up to 2 years.
  The rate of recruitment will be calculated as the number of months from the date of commencing recruitment to the date of randomizing the tenth participant.
Participant withdrawal rate, calculated as the number of participants who withdraw from the trial as a proportion of the total number of participants randomized. | Day 1 to day 176 (end of treatment period 2)
  The number of participants who withdraw from the trial will be calculated as a proportion of the total number of participants randomized.
Study medication tolerability, as indicated by the proportion of participants who tolerate the protocol dosing schedule. | Day 1 to day 176 (end of treatment period 2)
  The number of participants who adhere to the protocol dosing schedule without medication related protocol deviations, treatment discontinuations or dose modifications will be calculated as a proportion of the total sample for each treatment condition (medicinal cannabis or placebo).
Participant adherence to the study medication dosing schedule, calculated as the proportion of participants who demonstrate acceptable medication compliance. | Day 78 (end of treatment period 1) and day 176 (end of treatment period 2)
  Medication compliance will be assessed through pharmacy calculations from returned bottle volumes. Acceptable compliance will fall within the range of 80-120%. The number of participants with acceptable medication compliance will be reported as a proportion of the total sample randomized.
Study visit attendance, calculated as the proportion of visits completed across the study sample. | Screening to day 169 (final study visit)
  The number of study visits attended by all participants will be calculated as a proportion of the total possible visits in accordance with the study protocol.
Blood test completion, calculated as the proportion of blood tests completed across the study sample. | Screening to day 169 (final study visit)
  The number of study blood tests completed by all participants will be calculated as a proportion of the total possible blood tests in accordance with the study protocol.
Parent questionnaire completion, calculated as the proportion of parent-report questionnaires completed across the study sample. | Screening to day 169 (final study visit)
  The number of study questionnaires completed by all parents will be calculated as a proportion of the total possible questionnaires requiring completion in accordance with the study protocol.
Self-report questionnaire completion, calculated as the proportion of adolescent self-report questionnaires completed across the study sample. | Screening to day 169 (final study visit)
  The number of study self-report questionnaires completed by all participants will be calculated as a proportion of the total possible questionnaires requiring completion in accordance with the study protocol.
Study design acceptability will be evaluated through a parent-completed study specific evaluation questionnaire completed at the end of the study. | Day 197
  Study design acceptability will be assessed using an evaluation questionnaire developed specifically for this study, which uses Likert scales to assess satisfaction with recruitment, medication tolerability, frequency of study visits, burden of completing questionnaires, and overall study quality. Parents will complete this questionnaire at the end of their study participation (day 197). Data will be reported for each item individually, as the proportion of parents who responded positively on the Likert scale, where higher scores indicate more favorable responses.

SECONDARY OUTCOMES:
The frequency of adverse events as reported on the modified version of the Liverpool Adverse Event Profile (LAEP) at day 71 and day 169 will be summarized across the medicinal cannabis and placebo treatment phases. | Day 71 and 176
  Completed by the parent or guardian, the LAEP was designed to capture known side-effects of anti-epileptic medication. The modified version includes additional items to ascertain other known side-effects of medicinal cannabis. This measure includes 34 items. Adverse Events (AEs) reported on the LAEP will be considered significant if a 2-point increase in severity is reported from baseline to end of the maintenance dosing period (day 71 and day 176). The frequency of AEs meeting this criteria will be presented for the medicinal cannabis and placebo treatment phases respectively.
The frequency of adverse events as reported throughout the study will be summarized across the medicinal cannabis and placebo treatment phases. | Day 1 to day 197
  All possible adverse events will be recorded, as reported at study visits, during safety check phone calls and in between scheduled appointments. All Serious Adverse Events will be published, as well as all non-serious adverse events deemed by the investigators to be at least possibly related to the study drug. The frequency of these adverse events will be presented for the medicinal cannabis and placebo treatment phases respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Children's Hospital / Murdoch Children's Research Institute, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set collected for this analysis of the MC in TS Pilot Study will be available six months after publication of the primary outcome. The study protocol and analysis plan will also be available. The data must be obtained from the Murdoch Children's Research Institute. Prior to releasing any data the following are required: a data access agreement must be signed between relevant parties, the 'MC in TS Pilot Study' Study Management Group must see and approve the data analysis plan describing how the data will be analysed, there must be an agreement around appropriate acknowledgment and any additional costs involved must be covered. Should the Study Management Group be unavailable, this role is delegated to the Murdoch Children's Research Institute. Data will only be shared with a recognized research organisation which has approved the proposed analysis plan.
Supporting Information: Study Protocol, SAP
Time Frame: 6 months after publication of primary outcome
Access Criteria: 1) Data access agreement; 2) approval by Trial Steering Committee; 3) recognized research institutions.